CLINICAL TRIAL: NCT05028738
Title: Patient-oriented Randomized Pragmatic Feasibility Trial with RTMS in Depression and Anxiety
Acronym: PORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Fidel Vila-Rodriguez, MD, PhD, FRCPC, DFAPA, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H17-00161
Record Dates: First submitted 2021-08-07; First posted 2021-08-31 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Episode; Major Depressive Disorder
Keywords: Pragmatic; Patient-oriented research; TMS; Treatment-resistant depression; Transcranial Magnetic Stimulation; rTMS
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Two-arm, randomized feasibility trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single-masked (i.e. raters)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intermittent Theta Burst Stimulation (iTBS) (Active Comparator): iTBS to the L-DLPFC
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Low Frequency Right (LFR) (Active Comparator): 1Hz stimulation to the R-DLPFC
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — rTMS will employ the MagPro X100 stimulator equipped with the cool-B70 coil (MagVenture, Farum, Denmark). The dose will be a 120% resting motor threshold (rMT) in accordance to our latest trial using iTBS. Localization of the right and left DLPFC will follow the well-established Beam F3 procedure. Subjects will then undergo 30 sessions of rTMS, once daily on weekdays for 6 weeks. FDA-approved iTBS protocol will consist of bursts of 3 pulses at 50 Hz, bursts repeated at 5 Hz for 600 pulses total, 2 s on, 8 s off, for 3 min 9 sec, at 120% rMT. LFR will consist of 1 Hz stimulation consisting of a single train of 10min duration for 600 pulses total at 120% rMT.

SUMMARY:
This trial compares intermittent theta-burst stimulation (iTBS) to low frequency repetitive transcranial magnetic stimulation (LFR) in regards to depression and anxiety outcomes in 100 patients with treatment resistant depression (TRD).

DETAILED DESCRIPTION:
The overarching goal of this trial is to evaluate whether a definite adaptive pragmatic trial would be feasible and establish clear go/no-go criteria as to whether proceeding to such definite trial is feasible. Specific aims include 1) testing the feasibility of recruiting a sample of TRD patients with less strict inclusion and exclusion criteria; 2) comparing different depression and anxiety scales (both clinician-rated and self-rated) and seek input from patients regarding their preferences; 3) seek input from patients with regards to the use of digital phenotyping as a tool to investigate biomarkers as well as engaging in the design of a potential implementation of such biomarker in a future definite trial.

Aim 1. To evaluate the feasibility of a future definite adaptive pragmatic RCT comparing left vs right DLPFC repetitive transcranial magnetic stimulation (rTMS) in TRD.

Hypothesis 1a: Enrollment will be 70% of the planned target over the 1-year recruitment period.

Hypothesis 1b: Retention rate of randomized participants will be ≥70% at the end of the intervention in both groups.

Aim 2. To evaluate patients' preferences regarding information about treatment options when there is no response to allocated treatment.

Hypothesis 2: Patients will prefer to modify treatment when there is no response.

Aim 3. To assess the feasibility of digital phenotyping as an tool to investigate biomarkers in TRD.

Hypothesis 3a: Survey uptake and participation in the study regarding the use of digital phenotyping will be 80% of randomized participants. Hypothesis 3b: Of those survey responders, 75% will indicate they would consent to digital phenotyping in a future definite RCT.

Aim 4. To develop a Bayesian statistical model that continuously updates personalized treatment effect estimates as the trial progresses, and identify the circumstances under which use of the model in a full-scale trial could inform treatment choice as the trial progresses.

Hypothesis 4: The modeling results will identify at least one subgroup for whom early stopping of the definitive trial in that subgroup may be warranted.

ELIGIBILITY:
Inclusion Criteria:

1. are outpatients;
2. are voluntary and competent to consent to treatment;
3. are ≥ 18 years;
4. have a score ≥ 26 on the IDS-30-SR;
5. have had no increase or initiation of any psychotropic medication in the 4 weeks prior to screening;
6. able to adhere to the treatment schedule;
7. pass the TMS adult safety screening (TASS) questionnaire

Exclusion Criteria:

1. have active suicidal intent;
2. are pregnant;
3. have a lifetime diagnosis of schizophrenia, bipolar disorder type I, schizophreniform, schizoaffective disorder or presence of psychotic symptoms within last 3 months;
4. have a concomitant major unstable medical illness;
5. have any significant form of dementia or any history of epilepsy;
6. have any intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed;
7. If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study;
8. If they are taking psychotropic medication, be on a stable dose for 4 weeks before starting treatment, and no initiation of new regular psychotropic medication;
9. have a clinically significant laboratory abnormality, in the opinion of the one of the principal investigators;
10. have a non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Depression severity | one week post treatment
  Inventory of Depressive Symptoms (IDS-30-SR); Minimum value per question: 0; Maximum value per question: 3; Total minimum value: 0; Total maximum value: 84; Higher score means worse outcome.

SECONDARY OUTCOMES:
Suicidal ideation | one week post treatment
  Columbia-Suicide Severity Rating Scale (C-SSRS); This questionnaire has binary responses (Yes/No). More responses with "Yes" mean worse outcome.
Anxiety severity | one week post treatment
  Brief Symptom Inventory anxiety subscale (BSI-Anxiety); Minimum value per question: 0 (Not at all); Maximum value per question: 4 (Extremely); Total minimum value: 0; Total maximum value: 24; Higher score means worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Fidel Vila-Rodriguez, MD, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Non-Invasive Neurostimulation Therapies (NINET) Laboratory, UBC Department of Psychiatry, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No